CLINICAL TRIAL: NCT00071773
Title: A Pilot Study of Laser Photocoagulation for Diabetic Macular Edema
Acronym: Laser
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research (DRCR.net)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-113; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2003-10-30; First posted 2003-11-03 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; laser photocoagulation; etdrs; macular grid photocoagulation; DME

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Early Treatment Diabetic Retinopathy Study (ETDRS) (Active Comparator): modified-ETDRS
  Interventions: Procedure: modified-ETDRS photocoagulation
- Mild Macular Grid (MMG) (Active Comparator): MMG technique
  Interventions: Procedure: Mild Macular Grid photocoagulation

INTERVENTIONS:
Procedure: modified-ETDRS photocoagulation — A treatment session can be given in single or multiple sittings at the investigator's discretion, as long as the entire treatment session is completed within 6 weeks. Retreatment in Phase 1 of the study should only occur at the 3.5 and 8 month visits.
  Other Names: focal/grid photocoagulation
  Arms: Modified Early Treatment Diabetic Retinopathy Study (ETDRS)
Procedure: Mild Macular Grid photocoagulation — A treatment session can be given in single or multiple sittings at the investigator's discretion, as long as the entire treatment session is completed within 6 weeks. Retreatment in Phase 1 of the study should only occur at the 3.5 and 8 month visits.
  Other Names: mmg photocoagulation
  Arms: Mild Macular Grid (MMG)

SUMMARY:
This pilot study will compare the use of current laser treatment for diabetic macular edema with a similar laser treatment that is milder in intensity, but more extensive.

DETAILED DESCRIPTION:
Diabetic retinopathy is a disorder of major public health importance, accounting for the majority of visual loss among working age Americans. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20 percent in patients with type 1 diabetes mellitus (DM), 25 in patients with type 2 DM who are taking insulin, and 14 percent in patients with type 2 DM who do not take insulin. The Early Treatment Diabetic Retinopathy Study (ETDRS) showed that moderate vision loss, defined as a doubling of the visual angle (e.g., 20/20 reduced to 20/40), can be reduced by 50 percent or more by focal/grid laser photocoagulation according to ETDRS protocol. Although several treatment modalities are currently under investigation, the only demonstrated means to reduce the risk of vision loss from diabetic macular edema are ETDRS laser photocoagulation, as demonstrated by the ETDRS, and intensive glycemic control, as demonstrated by the Diabetes Control and Complications Trial (DCCT) and the United Kingdom Prospective Diabetes Study (UKPDS). In the DCCT, intensive glucose control reduced the risk of onset of diabetic macular edema by 23 percent compared with conventional treatment. Long-term follow-up of patients in the DCCT show a sustained effect of intensive glucose control, with a 58 percent risk reduction in the development of diabetic macular edema for the DCCT patients followed in the Epidemiology of Diabetes Interventions and Complications Study.

In brief, the study protocol involves the enrollment of patients >18 years of age who have DME involving or threatening the center of the macula and who have not had prior focal/grid laser photocoagulation for DME. These are patients for whom the standard of care would be to treat with laser photocoagulation. Eligible eyes will be randomly assigned to receive either the modified-ETDRS technique or the mild macular grid (MMG) technique. Outcome assessments will include Optical Coherence Tomography (OCT), fundus photography, fluorescein angiography and standardized best-corrected visual acuity.

The study consists of two phases: Phase 1 (the primary study), which consists of the first 12 months of follow up, during which a structured protocol is followed; and Phase 2, which consists of the second and third years of follow up, during which the management of DME can include techniques other than laser photocoagulation, at discretion of the investigator.

During Phase 1, follow-up visits will occur at 15 weeks (3.5 months) +14 days, 34 weeks (8 months) + 28 days, and 52 weeks (12 months) + 28 days. The primary outcome for phase 1 is at 12 months.

The primary study objectives of Phase 1 include:

* Develop standardized study procedures for future DME studies
* Obtain outcome data (e.g. changes in retinal thickness, area of retinal thickening, area of hard exudate, need for retreatment, onset of new areas of DME and changes in visual acuity) following use of the modified-ETDRS photocoagulation technique for patients with DME and various levels of retinopathy severity.
* Collect pilot data using the MMG technique to determine whether a subsequent large scale definitive trial should be conducted

Phase 2 (2nd and 3rd years of follow up) is being conducted to collect data on, and generate hypotheses from, the long-term outcome of DME, irrespective of treatment received. Protocol visits will occur at 2 years + 8 weeks and 3 years + 8 weeks. During this phase of the study, therapies other than laser photocoagulation may be used to treat DME at the investigator's discretion. Because treatment other than photocoagulation will be allowed after one year, 'pure' results regarding outcomes with each laser technique cannot be obtained in all groups, but will be available in a subset of patients. The data are being collected at relatively low cost and no risk over and above usual care. Therefore, the collection of potentially hypothesis-generating data from exploratory analysis is justified and could be important in designing future studies. Interpretation of the results of the above analyses will be complicated by the lack of a standardized protocol with regard to which patients receive treatment and what treatment is provided. Therefore, the results will be interpreted with caution.

The phase 2 data collection may be useful for the following:

* Evaluation of retreatment rates in patients who responded to laser such that no additional treatment was required at 12 months. This is a long term analysis on a "pure" group of patients and will provide important information on the DME recurrence rate and need for retreatment in study eyes of those patients whose DME improved with either of the two protocol-specified treatments received in Phase 1 such that further treatment was not necessary at the 12-month visit.
* Provide long-term safety data for MMG. This is important due to the less well studied nature of MMG, especially over the long term.
* Provide long-term outcome data on current standard treatment (modified ETDRS laser) in today's patient populations to assist in powering future studies that will require at least 3 years of follow up.
* Provide data on outcome of intravitreal steroids in patients in whom laser treatment is not successful. For many patients who still have DME at 12 months, it is anticipated that intravitreal steroids will be administered. The continued follow up of these patients will provide an opportunity to explore the effect of the steroids on retinal thickness and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years. Patients <18 years old are not being included because diabetic macular edema (DME) is so rare in this age group that the diagnosis of DME may be questionable.
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Any one of the following will be considered to be sufficient evidence that diabetes is present:

Current regular use of insulin for the treatment of diabetes; Current regular use of oral antihyperglycemia agents for the treatment of diabetes; Documented diabetes by ADA guidelines (see DRCR.net Procedures Manual).

* No history of renal failure requiring dialysis or renal transplant.
* No condition that in the opinion of the investigator would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control; Patients in poor glycemic control who recently initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 3 months should not be enrolled.
* Ability and willingness to provide informed consent.
* No expectation that subject will be moving out of the area of the clinical center to an area not covered by another clinical center during the next 12 months.

Study Eye Criteria:

At least one eye must meet all of the following criteria:

* Best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score >= 19 letters (approximately 20/400 or better).
* Definite retinal thickening due to diabetic macular edema based on clinical exam at or within 500 microns of the macular center for which the investigator believes laser photocoagulation is indicated.
* A thickness of 250 microns or more in the central subfield OR a thickness of 300 microns or more in any one of the four subfields directly adjacent to the central subfield on optical coherence tomography (OCT).
* No prior focal/grid laser photocoagulation in the macula.
* No prior medical treatment for DME (e.g., intravitreal/peribulbar steroids).
* No panretinal scatter photocoagulation (PRP) within prior 4 months.
* No anticipated need for PRP within next 4 months.
* No major ocular surgery (including cataract extraction, any other intraocular surgery, scleral buckle, glaucoma filter, cornea transplant, etc.) within prior 6 months.
* No Nd:YAG laser capsulotomy within prior 2 months.
* Macular edema is not considered to be due to a cause other than diabetic macular edema. An eye should not be considered eligible (1) if the macular edema is considered to be related to cataract extraction or (2) clinical exam and/or OCT suggests that vitreoretinal interface disease (eg. vitreo-retinal traction or epriretinal membrane) is the primary cause of the macular edema.
* Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photos.
* No ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the first 12 months of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome).
* Glaucoma per se is not an exclusion.

A patient may have two "study eyes" only if both are eligible at the time of randomization. An eye that becomes eligible after randomization will not be considered a study eye for purposes of data analyses or treatment decisions although information is being gathered on all eyes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2003-07; Primary Completion 2005-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in the central subfield of the ETDRS grid measured by OCT. | 1 Year

SECONDARY OUTCOMES:
Change in visual acuity | 1 Year
Change in area of retinal thickening on fundus photographs | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Donald S. Fong, MD, PhD, Study Chair — Kaiser Permanente

REFERENCES:
- [Result] Diabetic Retinopathy Clinical Research Network; Browning DJ, Glassman AR, Aiello LP, Beck RW, Brown DM, Fong DS, Bressler NM, Danis RP, Kinyoun JL, Nguyen QD, Bhavsar AR, Gottlieb J, Pieramici DJ, Rauser ME, Apte RS, Lim JI, Miskala PH. Relationship between optical coherence tomography-measured central retinal thickness and visual acuity in diabetic macular edema. Ophthalmology. 2007 Mar;114(3):525-36. doi: 10.1016/j.ophtha.2006.06.052. Epub 2006 Nov 21. PMID 17123615
- [Result] Davis MD, Bressler SB, Aiello LP, Bressler NM, Browning DJ, Flaxel CJ, Fong DS, Foster WJ, Glassman AR, Hartnett ME, Kollman C, Li HK, Qin H, Scott IU; Diabetic Retinopathy Clinical Research Network Study Group. Comparison of time-domain OCT and fundus photographic assessments of retinal thickening in eyes with diabetic macular edema. Invest Ophthalmol Vis Sci. 2008 May;49(5):1745-52. doi: 10.1167/iovs.07-1257. Epub 2008 Mar 3. PMID 18316700
- [Result] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Fong DS, Strauber SF, Aiello LP, Beck RW, Callanan DG, Danis RP, Davis MD, Feman SS, Ferris F, Friedman SM, Garcia CA, Glassman AR, Han DP, Le D, Kollman C, Lauer AK, Recchia FM, Solomon SD. Comparison of the modified Early Treatment Diabetic Retinopathy Study and mild macular grid laser photocoagulation strategies for diabetic macular edema. Arch Ophthalmol. 2007 Apr;125(4):469-80. doi: 10.1001/archopht.125.4.469. PMID 17420366
- [Result] Browning DJ, Apte RS, Bressler SB, Chalam KV, Danis RP, Davis MD, Kollman C, Qin H, Sadda S, Scott IU; Diabetic Retinopathy Clinical Research Network. Association of the extent of diabetic macular edema as assessed by optical coherence tomography with visual acuity and retinal outcome variables. Retina. 2009 Mar;29(3):300-5. doi: 10.1097/IAE.0b013e318194995d. PMID 19174719
- [Result] Scott IU, Danis RP, Bressler SB, Bressler NM, Browning DJ, Qin H; Diabetic Retinopathy Clinical Research Network. Effect of focal/grid photocoagulation on visual acuity and retinal thickening in eyes with non-center-involved diabetic macular edema. Retina. 2009 May;29(5):613-7. doi: 10.1097/IAE.0b013e3181a2c07a. PMID 19373126